CLINICAL TRIAL: NCT07220343
Title: Using Digital Phenotyping to Optimize Psychosocial Risk Screening and Personalized Care: a Pilot Study in Adolescents and Young Adults With Cancer
Brief Title: Digital Phenotyping for Psychosocial Screening in Adolescents and Young Adults With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-73748
Record Dates: First submitted 2025-09-09; First posted 2025-10-23 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Cancer; Adolescents
Keywords: Smartphone; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Equipment and Supplies; Ecological Momentary Assessment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital Phenotyping Arm (Experimental): All participants (adolescents and young adults with cancer) will receive the digital phenotyping intervention, which includes wearing a smartwatch and using a smartphone-based EMA app over a 10-day period, with psychosocial assessments at baseline, day 10, and 2 months
  Interventions: Device: Device; Behavioral: Ecological Momentary Assessment (EMA) via My Personal Health Dashboard (MyPHD) Smartphone App

INTERVENTIONS:
Device: Device — Participants will wear a wrist-based wearable device for 10 days to passively track physiological data (heart rate, steps, sleep, etc.).
Behavioral: Ecological Momentary Assessment (EMA) via My Personal Health Dashboard (MyPHD) Smartphone App — Participants will respond to ecological momentary assessments (EMA) via smartphone to actively report on sleep, mood, stress, and eating habits across a 10-day period.

SUMMARY:
The overall goal of the proposed study is to use digital phenotyping to identify and triage at-risk patients and accelerate access to critical mental health services.

ELIGIBILITY:
Inclusion Criteria:

* 10-25 years old
* Recent cancer diagnosis (>2 and <18 months since diagnosis)
* Willing to carry smartphone on their person for duration of study participation
* Willing to wear smartwatch for duration of study participation

Exclusion Criteria:

* Significant physical or mental disability that prevents completion of study activities
* Lack of proficiency in English or Spanish

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Depressive Symptoms (Beck Depression Inventory - BDI) | Baseline, Day 10, 2 months
  The Beck Depression Inventory-II (BDI-II; range 0-63) will be used to measure changes in depressive symptoms among adolescents and young adults over time. Higher scores indicate greater depressive symptom severity.

SECONDARY OUTCOMES:
Participant Retention Rate (MyPHD App and Wearable Device) | Baseline to 2 months
  Percentage of participants who remain active in the study through the 2-month follow-up period using the MyPHD app and wearable device.
Adherence to EMA Prompts | Baseline to 2 months
  Mean percentage of EMA prompts completed by participants using the MyPHD mobile app during the 2-month study period. Completion will be assessed via EMA system analytics.
Wearable Device Return and Use Rate | Baseline to 2 months
  Percentage of participants who return and use the wearable device as instructed during the study period. Device use will be tracked through backend device usage logs.
Change in Anxiety Symptoms (Beck Anxiety Inventory - BAI) | Baseline, Day 10, 2 months
  Measures changes in self-reported anxiety symptoms across the study period.
Change in PTSD Symptoms (CROPS) | Baseline
  PTSD symptoms are measured using the Child Report of Post-traumatic Symptoms (CROPS) for child participants.
Change in PTSD Symptoms (PCL-5) | Baseline
  PTSD symptoms are measured using the PTSD Checklist for DSM-5 (PCL-5) for general population participants.
Change in Sleep Quality (Pittsburgh Sleep Quality Index - PSQI) | Baseline, Day 10
  Assesses subjective sleep quality and patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Cosgrove, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States